CLINICAL TRIAL: NCT07277101
Title: Sensory-friendly Physical Activity and Sleep in Autistic Children: A Randomized Controlled Trial
Brief Title: Sensory-Friendly Physical Activity for Sleep in Autistic Children
Acronym: SFPAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xili Wen (Other)
Responsible Party: Sponsor-Investigator, Xili Wen, Principal Investigator, School of Physical Education and Training, Shanghai University of Sport, Shanghai University of Sport
Organization: Shanghai University of Sport (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUS-APA-ASD-SLEEP-RCT; SUS (Other: Shanghai University of Sport)
Record Dates: First submitted 2025-11-30; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Autism Spectrum Disorder; Sleep Initiation and Maintenance Disorders
Keywords: autism; autistic children; sleep problems; insomnia; sensory-friendly physical activity; school-based intervention; exercise program; randomized trial; actigraphy
MeSH Terms: conditions — Autism Spectrum Disorder; Sleep Initiation and Maintenance Disorders; Autistic Disorder; Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAP (Experimental): Classrooms receive a teacher-led, sensory-friendly physical activity program integrated into regular physical education lessons, 3 times per week for 16 weeks. Sessions include structured warm-up, adapted multi-component activities, and calming cool-down with breathing and relaxation in a low-arousal environment.
  Interventions: Behavioral: Sensory-Friendly Physical Activity Program (PAP)
- CC (Active Comparator): Classrooms continue usual school routines
  Interventions: Other: Conventional control group

INTERVENTIONS:
Behavioral: Sensory-Friendly Physical Activity Program (PAP) — A structured, teacher-led physical activity program designed to be sensory-friendly for autistic children. Delivered in special education schools during scheduled physical education lessons, 3 sessions per week for 16 weeks. Each session includes predictable routines, warm-up, moderate-to-vigorous activities adapted for motor and sensory needs, and a cool-down with breathing and relaxation to support self-regulation and sleep readiness.
  Arms: PAP
Other: Conventional control group — Children follow the usual daily schedule
  Arms: CC

SUMMARY:
Sleep problems are very common in children on the autism spectrum and can worsen daytime behaviour, learning, and family stress. Many families have limited access to specialist sleep services. This study evaluates a school-based, sensory-friendly physical activity program designed to improve sleep and wellbeing in autistic children.

This multicenter, parallel-group, cluster-randomized controlled trial was conducted in special education schools in China. Classrooms of children aged 7-12 years with a diagnosis of autism spectrum disorder were randomly assigned to either: (1) a teacher-led, sensory-friendly physical activity program integrated into regular physical education lessons for 16 weeks, or (2) usual school activities without the program. The intervention emphasized predictable routines, gradual warm-up, adjusted sensory input (for example, noise and light), and calming cool-down activities to support self-regulation and readiness for sleep.

The primary outcomes are children's sleep parameters measured by wrist actigraphy, including sleep efficiency, sleep onset latency, sleep duration, and wake after sleep onset. Secondary outcomes include parent-reported sleep problems, children's daily moderate-to-vigorous physical activity, and caregivers' sleep quality, mental health, parenting sense of competence, and quality of life. Outcomes are assessed at baseline, immediately after the 16-week program, and 6 months after the program ends.

DETAILED DESCRIPTION:
This study is a multicenter, parallel-group, cluster-randomized controlled trial conducted in special education schools in China. Classrooms are the unit of randomization to minimize contamination between children in the same class. Eligible participants are children aged 7-12 years with a documented diagnosis of autism spectrum disorder who attend participating special schools, have at least one sleep difficulty (such as bedtime resistance, prolonged sleep onset, or night wakings), and live with a primary caregiver who can complete questionnaires in Mandarin and provide informed consent.

Classes are randomly assigned in a 1:1 ratio to either the sensory-friendly Physical Activity Program (PAP) or a control condition. The PAP is delivered by trained physical education teachers during scheduled lessons, three times per week for 16 weeks. Each session includes a structured warm-up, multi-component physical activities adapted for motor and sensory needs, and a cool-down segment with breathing and relaxation exercises in a low-arousal environment. Teachers receive manuals and on-site coaching to support fidelity. The control group follows usual school routines and physical education without the PAP.

The primary outcomes are actigraphy-derived sleep parameters: sleep efficiency, sleep onset latency, total sleep time, and wake after sleep onset. Secondary outcomes include accelerometer-measured daily physical activity; parent-reported sleep problems; and caregiver-reported sleep quality, anxiety and depressive symptoms, parenting sense of competence, and health-related quality of life. Data are collected at three time points: baseline (before randomization), immediately after the 16-week intervention, and 6-month follow-up. Linear mixed-effects models with random intercepts for classroom and child are used to estimate intervention effects while accounting for clustering and prespecified covariates.

ELIGIBILITY:
Eligibility criteria Child inclusion criteria(1) Aged 7-12 years with a documented DSM-5 diagnosis of autism spectrum disorder in school records.(2) Able to understand and execute two-step instructions, as confirmed by the classroom special-education teacher.(3) Parent-reported sleep problems on the Children's Sleep Habits Questionnaire (CSHQ), operationalised as ≥ 5 nights per week of bedtime resistance, sleep onset delay, or night wakings.

Caregiver inclusion criteria (1) Identified as the child's primary caregiver in daily life.(2) Fluent in Mandarin (speaking, listening, reading, and writing), as all intervention and assessments were conducted in Mandarin.(3) ≥ 18 years of age.(4) Provided written informed consent and agreed to random allocation.

Exclusion criteria

(1) Current or prior pharmacological or behavioural treatment specifically targeting sleep.(2) Medical conditions that preclude participation in physical activity (e.g., asthma, congenital heart disease).(3) Comorbid complex neurological disorders (e.g., epilepsy) or other medical/psychiatric conditions likely to interfere with sleep.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Sleep Efficiency (SE) | Baseline (T0), post-intervention at 16 weeks (T1), and 6-month follow-up (T2).
  Actigraphy-derived sleep efficiency, calculated as (total sleep time / time in bed) × 100%, averaged across at least 3 consecutive nights at each assessment. Higher scores indicate more efficient sleep.
Sleep Onset Latency (SOL) | Baseline (T0), post-intervention at 16 weeks (T1), and 6-month follow-up (T2).
  Actigraphy-derived sleep onset latency, defined as the number of minutes from lights out (bedtime) to the onset of sustained sleep, averaged across at least 3 consecutive nights at each assessment. Lower scores indicate faster sleep initiation.
Total Sleep Time (TST) | Baseline (T0), post-intervention at 16 weeks (T1), and 6-month follow-up (T2).
  Actigraphy-derived total sleep time, defined as the total number of minutes scored as sleep between sleep onset and final morning waking, averaged across at least 3 consecutive nights at each assessment. Higher scores indicate longer nocturnal sleep duration.
Wake After Sleep Onset (WASO) | Baseline (T0), post-intervention at 16 weeks (T1), and 6-month follow-up (T2).
  Actigraphy-derived wake after sleep onset, defined as the cumulative number of minutes scored as wake after initial sleep onset until final morning waking, averaged across at least 3 consecutive nights at each assessment. Lower scores indicate less fragmented sleep.

SECONDARY OUTCOMES:
Daily Moderate-to-Vigorous Physical Activity (MVPA) | Baseline (T0), post-intervention at 16 weeks (T1), and 6-month follow-up (T2).
  Accelerometer-measured daily minutes of moderate-to-vigorous physical activity (MVPA). Children wear a wrist-worn accelerometer for 7 consecutive days at each assessment. Days with at least 10 hours of valid wear time are retained, and the average daily MVPA minutes are calculated. Higher values indicate greater physical activity.
Parental Sleep Quality (PSQI Total Score) | Baseline (T0), post-intervention at 16 weeks (T1), and 6-month follow-up (T2).
  Caregiver-reported global sleep quality measured by the Pittsburgh Sleep Quality Index (PSQI). The PSQI yields a total score ranging from 0 to 21, with higher scores indicating poorer sleep quality.
Parenting Sense of Competence (PSOC Total Score) | Baseline (T0), post-intervention at 16 weeks (T1), and 6-month follow-up (T2).
  The PSOC has 16 items rated on a 6-point Likert scale, yielding a total score from 16 to 96; higher scores indicate greater parenting sense of competence.
Caregiver Anxiety Symptoms (HADS-A Subscale Score) | Baseline (T0), post-intervention at 16 weeks (T1), and 6-month follow-up (T2).
  Caregiver anxiety symptoms measured by the Anxiety subscale of the Hospital Anxiety and Depression Scale (HADS-A). The subscale comprises 7 items scored 0-3, yielding a total score from 0 to 21, with higher scores indicating more severe anxiety symptoms.
Caregiver Depressive Symptoms (HADS-D Subscale Score) | Baseline (T0), post-intervention at 16 weeks (T1), and 6-month follow-up (T2).
  Caregiver depressive symptoms measured by the Depression subscale of the Hospital Anxiety and Depression Scale (HADS-D). The subscale comprises 7 items scored 0-3, yielding a total score from 0 to 21, with higher scores indicating more severe depressive symptoms.
Caregiver Health-Related Quality of Life (WHOQOL-BREF Domain Scores) | Baseline (T0), post-intervention at 16 weeks (T1), and 6-month follow-up (T2).
  Health-related quality of life measured by the World Health Organization Quality of Life-BREF (WHOQOL-BREF). The instrument yields four domain scores (Physical Health, Psychological Health, Social Relationships, and Environment). Domain scores are transformed to a 0-100 scale, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai University of Sport, School of Physical Education and Training, Shanghai, China